CLINICAL TRIAL: NCT02857660
Title: Effect of Whole-body Electromyostimulation (WB-EMS) and/or Protein Supplementation on Sarcopenic Obesity in Community Dwelling Males 70+ With Sarcopenic Obesity
Brief Title: Effect of Whole Body Electromyostimulation and/or Protein Supplementation on Sarcopenic Obesity in 70+
Acronym: FRANSO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: University of Erlangen-Nürnberg Institute of Medical Physics (Unknown); University of Erlangen-Nürnberg Institute of Biomedicine of Aging (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FRANSO_2016_IMP
Record Dates: First submitted 2016-07-28; First posted 2016-08-05 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Sarcopenic Obesity
Keywords: Sarcopenia; Obesity; Whole-Body Electromyostimulation; Protein Supplementation; community dwelling men
MeSH Terms: conditions — Sarcopenia; Obesity | interventions — Exercise; Transcutaneous Electric Nerve Stimulation; Proteins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Whole-Body Electromyostimulation and Protein (Experimental): 16 weeks of whole-body intervention 1.5 x 20 min week with bipolar current up to 1.5 - 1.7 g/kg body mass/d of protein supplements up to 800 IU/d Vitamin D-Supplementation
  Interventions: Other: Whole body Electromyostimulation (exercise); Dietary Supplement: Protein
- Protein supplementation (Active Comparator): up to 1.5 - 1.7 g/kg body mass/d of protein supplements up to 800 IU/d Vitamin D-Supplementation
  Interventions: Dietary Supplement: Protein
- sedentary Control Group (No Intervention): No protein supplementation or WB-EMS-application, but up to 800 IU/d Vitamin D-Supplementation

INTERVENTIONS:
Other: Whole body Electromyostimulation (exercise) — 1.5 x 20 min/week (e.g. each Tuesday and every second Friday) with bipolar current, 85 Hz, 360 µs, rectangular mode, intermittent with 4 sec of current and 4 s of rest.
  Other Names: Electrostimulation
  Arms: Whole-Body Electromyostimulation and Protein
Dietary Supplement: Protein — up to 1.5-1.7 g/kg bodymass/d of protein (whey protein)
  Arms: Protein supplementation; Whole-Body Electromyostimulation and Protein

SUMMARY:
The aim of the study is to determine the effect of 16 weeks of Whole Body-Electromyostimulation (WB-EMS) and/or protein supplementation on Sarcopenic Obesity (SO) in community dwelling male subjects 70+ with SO .

108 eligible men will be randomly assigned to either a (1) WB-EMS and Protein (2) Protein (3) sedentary control group.

WB-EMS will be applied 1,5 x 20 min per week (i.e. 3 sessions in two weeks) with bipolar current, 85 Hz in an intermitted mode (4 s - 4 s of rest). Protein supplementation will be adjusted to dietary intake in order to reach a total protein intake between 1,5 - 1,7g/kg body-mass/d . Primary study endpoint will be the Sarcopenia Z-Score

DETAILED DESCRIPTION:
The aim of the study is to evaluate the effects of Whole-Body Electromyostimulation (WB-EMS) with additional protein supplementation on Sarcopenic Obesity parameters in independently living men 70 years and older with sarcopenic obesity. The randomized controlled study compares three groups with 36 subjects each: (1) WB-EMS with additional protein supplementation, (2) protein-only and (3) passive control group, over a period of 16 weeks of WB-EMS -training. Group (1) conducts 1.5-times/week a 20 minute-sessions of WB-EMS with additional protein, group (2) is limited to protein supplementation (only) and group (3) is constrained to maintain their habitual living behavior and physical activity. Based on an individual nutrition analysis the protein intake will be adjusted to 1.5-1.7 g/kg/ bodymass/d. All groups will be supplemented with a maximum of 800 IE Vitamin D.

Primary study endpoint will be changes of the Sarcopenia Z-Score with skeletal muscle mass assessed via bio-impedance analysis (BIA). Secondary study endpoints are changes of Obesity (i.e. body-fat as assessed via BIA), cardiometabolic risk (i.e. Metabolic Syndrome Z-Score), strength parameters evaluated via Dr. Wolff BackCheck and Physiomed LegPress, quality of life (SF-12) and functional disability (late life physical disability index).

ELIGIBILITY:
Inclusion Criteria:

* community dwelling, independent living men
* Sarcopenia
* Obesity (body fat >=25%)

Exclusion Criteria:

* exclusion criteria for WB-EMS-application (e.g. cardiac pacemaker)
* diseases/medication that affect the study endpoints (e.g. Glucocorticoids >5mg/d)
* absence of more than 2 weeks during the study period

Min Age: 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change of Sarcopenia Z-Score | Change from Baseline Sarcopenia Z-Score at 16 weeks
  ie. Z-Score generated by skeletal muscle index, gait speed and grip-strength according to the Sarcopenia Definition of the European Working Group on Sarcopenia in Older People
Change of Obesity | Change from Baseline Obesity at 16 weeks
  Assessment of body fat content and body mass index

SECONDARY OUTCOMES:
Change of Metabolic Syndrome Z-Score | Change from Baseline Metabolic Syndrome Z-Score at 16 weeks
  Metabolic Syndrome according to the International Diabetes Federation (IDF)
Change of isokinetic leg strength | Change from Baseline isokinetic leg strength at 16 weeks
  Dynamic strength of the leg extensors and flexors as determined by a isokinetic leg press
Change of Quality of Life | Change from Baseline Quality of life at 16 weeks
  Quality of life as determined by the SF-12 questionnaire
Change of Physical Disability | Change from Baseline Physical Disability at 16 weeks
  Physical disability as assessed by Late Life Functional and Disability Index (LLFDI)
Change of Back Extensors Strength | Change from Baseline Back Extensors Strength at 16 weeks
  Strength of the back extensors and flexors using the Doctor Wolff Backcheck device

CONTACTS AND LOCATIONS:
Overall Officials: Cornel Sieber, MD, Study Chair — Institute of Biomedicine of Aging, University of Erlangen-Nürnberg; Klaus Engelke, PhD, Study Chair — University of Erlangen-Nürnberg Medical School; Ellen Freiberger, PhD, Study Chair — Institute of Biomedicine of Aging, University of Erlangen-Nürnberg; Anja Weissenfels, MA, Principal Investigator — University of Erlangen-Nürnberg Medical School; Wolfgang Kemmler, PhD, Study Director — University of Erlangen-Nürnberg Medical School
Locations (1):
- Institute of Medical Physics, Friedrich Alexander University Erlangen-Nürnberg, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kemmler W, Teschler M, Weissenfels A, Bebenek M, von Stengel S, Kohl M, Freiberger E, Goisser S, Jakob F, Sieber C, Engelke K. Whole-body electromyostimulation to fight sarcopenic obesity in community-dwelling older women at risk. Resultsof the randomized controlled FORMOsA-sarcopenic obesity study. Osteoporos Int. 2016 Nov;27(11):3261-3270. doi: 10.1007/s00198-016-3662-z. Epub 2016 Jun 12. PMID 27289534
- [Background] Kemmler W, Teschler M, Goisser S, Bebenek M, von Stengel S, Bollheimer LC, Sieber CC, Freiberger E. Prevalence of sarcopenia in Germany and the corresponding effect of osteoarthritis in females 70 years and older living in the community: results of the FORMoSA study. Clin Interv Aging. 2015 Oct 3;10:1565-73. doi: 10.2147/CIA.S89585. eCollection 2015. PMID 26491272
- [Background] Kemmler W, von Stengel S, Engelke K, Sieber C, Freiberger E. Prevalence of sarcopenic obesity in Germany using established definitions: Baseline data of the FORMOsA study. Osteoporos Int. 2016 Jan;27(1):275-81. doi: 10.1007/s00198-015-3303-y. Epub 2015 Aug 29. PMID 26318759
- [Background] Goisser S, Kemmler W, Porzel S, Volkert D, Sieber CC, Bollheimer LC, Freiberger E. Sarcopenic obesity and complex interventions with nutrition and exercise in community-dwelling older persons--a narrative review. Clin Interv Aging. 2015 Aug 6;10:1267-82. doi: 10.2147/CIA.S82454. eCollection 2015. PMID 26346071
- [Derived] Chaudry O, Friedberger A, Grimm A, Uder M, Nagel AM, Kemmler W, Engelke K. Segmentation of the fascia lata and reproducible quantification of intermuscular adipose tissue (IMAT) of the thigh. MAGMA. 2021 Jun;34(3):367-376. doi: 10.1007/s10334-020-00878-w. Epub 2020 Aug 6. PMID 32761398
- [Derived] Kemmler W, Grimm A, Bebenek M, Kohl M, von Stengel S. Effects of Combined Whole-Body Electromyostimulation and Protein Supplementation on Local and Overall Muscle/Fat Distribution in Older Men with Sarcopenic Obesity: The Randomized Controlled Franconia Sarcopenic Obesity (FranSO) Study. Calcif Tissue Int. 2018 Sep;103(3):266-277. doi: 10.1007/s00223-018-0424-2. Epub 2018 Apr 19. PMID 29675640
- [Derived] Kemmler W, Kohl M, Freiberger E, Sieber C, von Stengel S. Effect of whole-body electromyostimulation and / or protein supplementation on obesity and cardiometabolic risk in older men with sarcopenic obesity: the randomized controlled FranSO trial. BMC Geriatr. 2018 Mar 9;18(1):70. doi: 10.1186/s12877-018-0759-6. PMID 29523089
- [Derived] Kemmler W, Teschler M, Weissenfels A, Sieber C, Freiberger E, von Stengel S. Prevalence of sarcopenia and sarcopenic obesity in older German men using recognized definitions: high accordance but low overlap! Osteoporos Int. 2017 Jun;28(6):1881-1891. doi: 10.1007/s00198-017-3964-9. Epub 2017 Feb 20. PMID 28220197